CLINICAL TRIAL: NCT01384513
Title: A Two Step Approach to Reduced Intensity Allogeneic Hematopoietic Stem Cell Transplantation for Patients With Hematologic Malignancies
Brief Title: A Two-Step Approach to Reduced Intensity Bone Marrow Transplant for Patients With Hematological Malignancies
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Cancer Center at Thomas Jefferson University (Other)
Responsible Party: Sponsor
Organization: Thomas Jefferson University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11D.247; 2011-31 (Other: CCRRC)
Record Dates: First submitted 2011-06-27; First posted 2011-06-29 (Estimated); Last update posted 2022-11-17 (Actual); Status verified 2022-11

CONDITIONS: Adult Acute Lymphoblastic Leukemia in Remission; Adult Acute Myeloid Leukemia in Remission; Adult Acute Myeloid Leukemia With 11q23 (MLL) Abnormalities; Adult Acute Myeloid Leukemia With Del(5q); Adult Acute Myeloid Leukemia With Inv(16)(p13;q22); Adult Acute Myeloid Leukemia With t(15;17)(q22;q12); Adult Acute Myeloid Leukemia With t(16;16)(p13;q22); Adult Acute Myeloid Leukemia With t(8;21)(q22;q22); Adult Nasal Type Extranodal NK/T-cell Lymphoma; Aplastic Anemia; Childhood Acute Lymphoblastic Leukemia in Remission; Childhood Acute Myeloid Leukemia in Remission; Childhood Myelodysplastic Syndromes; Chronic Eosinophilic Leukemia; Chronic Myelomonocytic Leukemia; Chronic Neutrophilic Leukemia; Essential Thrombocythemia; Extranodal Marginal Zone B-cell Lymphoma of Mucosa-associated Lymphoid Tissue; Juvenile Myelomonocytic Leukemia; Mastocytosis; Myelodysplastic/Myeloproliferative Neoplasm, Unclassifiable; Nodal Marginal Zone B-cell Lymphoma; Polycythemia Vera; Previously Treated Myelodysplastic Syndromes; Primary Myelofibrosis; Recurrent Adult Acute Lymphoblastic Leukemia; Recurrent Adult Acute Myeloid Leukemia; Recurrent Adult Diffuse Small Cleaved Cell Lymphoma; Recurrent Adult Grade III Lymphomatoid Granulomatosis; Recurrent Adult Hodgkin Lymphoma; Recurrent Childhood Acute Lymphoblastic Leukemia; Recurrent Childhood Acute Myeloid Leukemia; Recurrent Cutaneous T-cell Non-Hodgkin Lymphoma; Recurrent Grade 1 Follicular Lymphoma; Recurrent Grade 2 Follicular Lymphoma; Recurrent Marginal Zone Lymphoma; Recurrent Mycosis Fungoides/Sezary Syndrome; Recurrent Small Lymphocytic Lymphoma; Recurrent/Refractory Childhood Hodgkin Lymphoma; Refractory Anemia; Refractory Anemia With Ringed Sideroblasts; Refractory Hairy Cell Leukemia; Refractory Multiple Myeloma; Secondary Myelodysplastic Syndromes; Splenic Marginal Zone Lymphoma; T-cell Large Granular Lymphocyte Leukemia; Waldenström Macroglobulinemia
Keywords: Allogeneic HSCT; Hematopoietic stem cell transplantation
MeSH Terms: conditions — Congenital Abnormalities; Lymphoma, Extranodal NK-T-Cell; Anemia, Aplastic; Pdgfra-Associated Chronic Eosinophilic Leukemia; Leukemia, Myelomonocytic, Chronic; Leukemia, Neutrophilic, Chronic; Thrombocythemia, Essential; Leukemia, Myelomonocytic, Juvenile; Mastocytosis; Myeloproliferative Disorders; Lymphoma, B-Cell, Marginal Zone; Polycythemia Vera; Primary Myelofibrosis; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Lymphoma, Non-Hodgkin; Hodgkin Disease; Lymphoma, T-Cell, Cutaneous; Lymphoma, Follicular; Mycosis Fungoides; Sezary Syndrome; Leukemia, Lymphocytic, Chronic, B-Cell; Recurrence; Anemia, Refractory; Leukemia, Hairy Cell; Multiple Myeloma; Leukemia, Large Granular Lymphocytic; Waldenstrom Macroglobulinemia | interventions — fludarabine; fludarabine phosphate; Busulfan; Whole-Body Irradiation; Radiotherapy; Cyclophosphamide; Tacrolimus; Mycophenolic Acid; Peripheral Blood Stem Cell Transplantation; Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Treatment (Allogeneic PBSCT) (Experimental): REDUCED INTENSITY CONDITIONING: Patients receive fludarabine phosphate IV over 60 minutes on days -11 to -8 and busulfan IV over 3 hours on days -10 to -9. Patients undergo TBI on day -6. Patients also receive cyclophosphamide IV over 2 hours on days -3 and -2.
  TRANSPLANTATION: Patients undergo DLI on day -6 and CD-34+ allogeneic PBSCT on day 0.
  GVHD PROPHYLAXIS: Beginning on day -1, patients receive tacrolimus IV or PO with taper beginning on day 42. Patients also receive mycophenolate mofetil IV BID on days -1 to 28.
  Interventions: Drug: Fludarabine; Drug: Busulfan; Radiation: Total Body Irradiation (TBI); Biological: Donor Lymphocyte Infusion (DLI); Drug: Cyclophosphamide (CY); Drug: Tacrolimus; Drug: Mycophenolate mofetil; Device: Allogeneic hematopoietic stem cell transplantation; Procedure: Peripheral blood stem cell transplantation (PBSCT)

INTERVENTIONS:
Drug: Fludarabine — Given IV
  Other Names: fludarabine phosphate; Fludara
Drug: Busulfan — Given IV
  Other Names: Myleran; Busulfex IV
Radiation: Total Body Irradiation (TBI) — 2 Gy administered as part of the conditioning regimen
  Other Names: radiotherapy
Biological: Donor Lymphocyte Infusion (DLI) — Undergo DLI
  Other Names: buffy coat fusion
Drug: Cyclophosphamide (CY) — Given IV
  Other Names: Endoxan; Cytoxan; Neosar; Procytox; Revimmune; cytophosphane
Drug: Tacrolimus — Given IV or PO
  Other Names: FK-506; Fujimycin
Drug: Mycophenolate mofetil — Given IV
  Other Names: MMF; CellCept
Device: Allogeneic hematopoietic stem cell transplantation — Undergo CD34+ allogeneic PBSCT
  Other Names: CliniMACS
Procedure: Peripheral blood stem cell transplantation (PBSCT) — Undergo CD34+ allogeneic PBSCT
  Other Names: PBPC transplantation; PBSC transplantation; peripheral blood progenitor cell transplantation; transplantation; peripheral blood stem cell

SUMMARY:
The purpose of this research study is to compare the survival rates of patients with better risk disease undergoing hematopoietic stem cell transplant (HSCT) to the survival rates reported in the medical literature of similar patients undergoing reduced intensity HSCT from matched related donors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To compare the overall survival (OS) rate at 2 years post treatment using the Jefferson 2 step reduced intensity conditioning (RIC) approach in patients with haploidentical family donors with hematological malignancies in morphological or radiographic remission or with chemosensitive, indolent diseases to historical OS rates in similar populations after RIC matched donor HSCT as reported in the literature.

SECONDARY OBJECTIVES:

I. To compare the treatment-related mortality (TRM) rate at 2 years for patients treated on this study to the historical TRM rates of patients undergoing RIC matched-sibling HSCT as reported in the literature.

II. To compare the 2 year relapse rates and relapse related mortality of patients with myeloid diseases to that of patients with lymphoid diseases who are treated on this Thomas Jefferson University (TJU) RIC 2 step approach.

III. To determine the incidence and severity of graft-versus-host disease (GVHD) in patients undergoing treated on the TJU RIC 2 step approach.

IV. To evaluate engraftment rates and lymphoid reconstitution in patients treated on the TJU RIC 2 step approach.

V. To evaluate the incidence of TRM at 100 days in patients treated on the TJU RIC 2 step approach.

OUTLINE:

REDUCED INTENSITY CONDITIONING: Patients receive fludarabine phosphate intravenously (IV) over 60 minutes on days -11 to -8 and bulsufan IV over 3 hours on days -10 to -9. Patients undergo total body irradiation (TBI) on day -6. Patients also receive cyclophosphamide IV over 2 hours on days -3 and -2.

TRANSPLANTATION: Patients undergo donor lymphocyte infusion (DLI) on day -6 and cluster of differentiation (CD)-34+ allogeneic peripheral blood stem cell transplantation (PBSCT) on day 0.

GVHD PROPHYLAXIS: Beginning on day -1, patients receive tacrolimus IV or orally (PO) with taper beginning on day 42. Patients also receive mycophenolate mofetil IV twice daily (BID) on days -1 to 28.

After completion of study treatment, patients are followed up periodically for 2 years.

ELIGIBILITY:
Inclusion Criteria:

1. Any patient with hematologic or oncologic diagnosis in which allogeneic HSCT is thought to be beneficial, and in whom front-line therapy has already been applied. Patients treated on this protocol will be without morphological evidence of disease (complete remission or "CR"), or if the patient has evidence of disease, the patient must have had at least a good partial response (PR) to the most recent therapy and the disease must be chemoresponsive.
2. Patients treated on this study will have:

   * Acute leukemia in 1st or 2nd CR
   * MDS (myelodysplastic syndrome), specific subtypes of RA (refractory anemia) or RARS (refractory anemia with ringed sideroblasts) subtypes.
   * Hodgkin or Indolent Non-Hodgkin's lymphoma with chemosensitive disease
   * Myeloma without morphological evidence of disease, or a deep PR to the most recent therapy
   * Myeloproliferative disorders with at least a PR to current therapy
   * Aplastic Anemia
   * A hematological or oncological disease (not listed) that meets the criteria reviewed above (in CR or with a good PR).
3. Patients must have a related donor who is HLA mismatched at 2, 3, or 4 antigens at the HLA-A; B; C; DR loci in the GVHD direction. (Patients with related donors who are HLA identical or are a 1-antigen mismatch may be treated on this therapeutic approach, but will have their outcomes will not be part of the statistical aims of the study (see Summary section).
4. Patients must adequate organ function:

   * LVEF (Left ventricular end diastolic function) of >50%
   * DLCO (Diffusing Capacity of the Lung for Carbon Monoxide ) ≥50% of predicted corrected for hemoglobin
   * Adequate liver function as defined by a serum bilirubin <1.8, AST or ALT < 2.5X upper limit of normal
   * Creatinine Clearance of ≥ 60 mL/min
5. Performance status ≥ 80% (TJU Karnofsky) for patients ≥ 60 years old or ≥70% for patients < 60 years old.
6. HCT-CI Score ≤ 4 points for patients ≥ 60 years old or ≤ 5 points for patients < 60 years old.
7. Patients must be willing to use contraception if they have childbearing potential
8. Able to give informed consent

Exclusion Criteria:

1. Performance status < 80% (TJU Karnofsky) for patients ≥ 60 years old or <70% for patients < 60.
2. Hematopoietic Cell Transplant-Comorbidity Index (HCT-CI) Score > 4 points for patients ≥ 60 years old or > 5 points for patients < 60.
3. HIV positive
4. Active involvement of the central nervous system with malignancy
5. Inability to obtain informed consent
6. Pregnancy
7. Patients with life expectancy of < 6 months for reasons other than their underlying hematologic/oncologic disorder
8. Patients who have received alemtuzumab within 8 weeks of the transplant admission, or who have recently received horse or rabbit anti-thymocyte globulin and have an anti-thymocyte globulin level of > 2 ugm/ml
9. Patients with evidence of another malignancy, exclusive of a skin cancer that requires only local treatment, should not be enrolled on this protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2011-08-04 (Actual); Primary Completion 2020-11-13 (Actual); Study Completion 2022-11-16 (Actual)

PRIMARY OUTCOMES:
Overall Survival (OS) in patients with haploidentical family donors with hematological malignancies in morphological or radiographic remission or with chemosensitive, indolent diseases | At 2 years
  The primary null hypothesis is that 2 year OS rate is at most 35%. This hypothesis will be rejected if the 95% confidence interval for year OS rate computed from the estimated Kaplan-Meier survival curves will be entirely above 0.35.

SECONDARY OUTCOMES:
Treatment Related Mortality (TRM) | At 2 years
  To compare the treatment related mortality rate (TRM) for patients treated on this study to the historical TRM rates of patients undergoing reduced intensity conditioning (RIC) matched-sibling hematopoietic stem cell transplant (HSCT) as reported in the literature
Incidence and severity of GVHD, graded according to standard criteria | Assessed up to 2 years
  The estimates of incidence rates will be presented with corresponding 95% confidence intervals using the exact method
Relapse Rate | At 2 years
  Evaluated by estimating Kaplan-Meier survival curves. From these curves, the 95% confidence interval for 2 year rates will be computed.
Engraftment Rates | Assessed up to 2 years
  The estimates of incidence rates will be presented with corresponding 95% confidence intervals using the exact method.
Incidence of Treatment Related Mortality (TRM) | At 100 days
  The estimates of incidence rates will be presented with corresponding 95% confidence intervals using the exact method.
Relapse Related Mortality | At 2 years
  Evaluated by estimating Kaplan-Meier survival curves. From these curves, the 95% confidence interval for 2 year rates will be computed.
Lymphoid Reconstitution | 100 days post-transplant
  To evaluate lymphoid reconstitution in patients treated on the Two Step approach

CONTACTS AND LOCATIONS:
Overall Officials: Dolores Grosso, DNP, CRNP, Principal Investigator — Sidney Kimmel Cancer Center at Thomas Jefferson University; Neal Flomenberg, MD, Principal Investigator — Sidney Kimmel Cancer Center at Thomas Jefferson University
Locations (1):
- Thomas Jefferson University, Philadelphia, Pennsylvania, United States

REFERENCES:
- See also: Kimmel Cancer Center at Thomas Jefferson University, an NCI-Designated Cancer Center — http://www.KimmelCancerCenter.org
- See also: Thomas Jefferson University Hospitals — http://www.JeffersonHospital.org